CLINICAL TRIAL: NCT05125835
Title: Long-Term Periodontal Outcomes in Males and Females Following Sanative Therapy or Regular Hygiene Appointments and COVID-19
Brief Title: Periodontal Maintenance and the COVID-19 Pandemic
Status: Completed | Type: Observational
Sponsor: Brock University (Other)
Collaborators: Dr. Peter C. Fritz, Periodontal Wellness & Implant Surgery (Other)
Responsible Party: Principal Investigator, Wendy E. Ward, Ph.D., Professor & Canada Research Chair, Brock University
Other Study IDs: 21-037
Record Dates: First submitted 2021-11-15; First posted 2021-11-18 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Periodontal Diseases; Periodontal Pocket
Keywords: Periodontal therapy; Periodontal maintenance; Hygiene appointment; Sanative therapy; COVID-19
MeSH Terms: conditions — Periodontal Diseases; Periodontal Pocket; COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Periodontal disease is a chronic condition affecting the teeth and surrounding support structures, characterized by tooth loss and alveolar bone loss. Sanative therapy (ST) is the gold standard non-surgical treatment for periodontal disease and involves mechanically removing the subgingival bacteria from the periodontal pockets. Regular periodontal maintenance appointments are needed to maintain periodontal health after ST. Moreover, the periodontal health of individuals not requiring ST is also dependent on regular hygiene appointments. Due to Ontario's March 2020 COVID-19-related clinic closure for approximately 3 months along with a reduced numbers of appointments available due to guidelines of professional bodies and public health beyond this period of time, many appointments were considerably delayed or cancelled. The effects of this disruption to periodontal health in male and female patients who have undergone ST and continue with maintenance appointments or who attend for regular hygiene appointments have not yet been investigated.

DETAILED DESCRIPTION:
Sanative therapy (ST) is often the first line of treatment following a diagnosis of periodontal disease. By mechanically removing the inflammation-inducing bacteria below the gum line, a more controlled state of periodontal health can be achieved. Improvements in periodontal health achieved through ST can be maintained long-term with regular maintenance appointments that aid in preventing further progression of the disease. However, due to the government-mandated clinic closure in March 2020 of dental offices for all but emergency in-person care in Canada due to the COVID-19 pandemic, clinics were shut down for approximately 3 months with a reduced availability of appointments in the following year due to professional guidelines. Regular hygiene appointments (cleanings) were also considerably delayed or cancelled. This disruption in routine care, accompanied with the potential exacerbation of various risk factors for periodontal disease such as stress, diet, physical activity, and smoking or alcohol use brought on by the pandemic has not yet been investigated pertaining to the effect on clinical periodontal outcomes. The main objective of this study is to determine if delays in regularly scheduled maintenance or regular hygiene appointments caused by COVID-19 impacted clinical periodontal outcomes in male and female patients. Secondary objectives include retrospectively determining the long-term clinical outcomes of patients who underwent periodontal therapy or who have had regular hygiene appointments at the clinic; comparing the long-term periodontal outcomes of patients who undergo maintenance appointments and those who receive only regular hygiene appointments; and examining whether there exists a sex-specific response to either treatment. Periodontal outcomes of interest include probing depth, bleeding on probing, plaque index, and tooth loss.

ELIGIBILITY:
Inclusion Criteria:

* Have undergone sanative therapy or attend regular hygiene appointments at the clinic
* Age 19 years or older
* Willing and able to provide informed consent

Exclusion Criteria:

* Age < 19 years
* Unable to provide informed consent

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who have undergone either sanative therapy plus at least one maintenance appointment or who attend regular hygiene appointments at this clinic.
Sampling Method: Non-Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2021-11-21 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Probing Depth | Pre-sanative therapy
  This is a routine clinical measure of periodontal health (measured in mm)
Probing Depth | 8-12 weeks post-sanative therapy
  This is a routine clinical measure of periodontal health (measured in mm)
Probing Depth | At maintenance appointment (present day) and retrospectively from the clinical record from first maintenance appointment after the 8-12 weeks post-sanative therapy
  This is a routine clinical measure of periodontal health (measured in mm) for patients who attend the clinic for maintenance appointments after sanative therapy
Probing Depth | At hygiene appointment (present day) and retrospectively from the clinical record from first hygiene appointment at clinic, up to 17 years previously
  This is a routine clinical measure of periodontal health (measured in mm) in patients who attend the clinic for regular hygiene appointments
Bleeding on Probing | Pre-sanative therapy
  This is a clinical measure of inflammation and represented as the percent of bleeding sites that are measured at 6 sites per tooth.
Bleeding on Probing | 8-12 weeks post-sanative therapy
  This is a clinical measure of inflammation and represented as the percent of bleeding sites that are measured at 6 sites per tooth.
Bleeding on Probing | At maintenance appointment (present day) and retrospectively from the clinical record from first maintenance appointment after the 8-12 weeks post-sanative therapy
  This is a clinical measure of inflammation and represented as the percent of bleeding sites that are measured at 6 sites per tooth.
Bleeding on Probing | At hygiene appointment (present day) and retrospectively from the clinical record from first hygiene appointment at clinic, up to 17 years previously
  This is a clinical measure of inflammation and represented as the percent of bleeding sites that are measured at 6 sites per tooth.

SECONDARY OUTCOMES:
O'Leary Index of Plaque Control | Pre-sanative therapy
  The patient's plaque index= the number of plaque-containing surfaces divided by the total number of available surfaces. The minimum plaque index would be 0% which represents no tooth surfaces that contain plaque/ The maximum plaque index would be 100%, which represents all surfaces of the patient's teeth containing plaque.
O'Leary Index of Plaque Control | 8-12 weeks post-sanative therapy
  The patient's plaque index= the number of plaque-containing surfaces divided by the total number of available surfaces. The minimum plaque index would be 0% which represents no tooth surfaces that contain plaque/ The maximum plaque index would be 100%, which represents all surfaces of the patient's teeth containing plaque.
O'Leary Index of Plaque Control | At maintenance appointment (present day) and retrospectively from the clinical record from first maintenance appointment after the 8-12 weeks post-sanative therapy
  The patient's plaque index= the number of plaque-containing surfaces divided by the total number of available surfaces. The minimum plaque index would be 0% which represents no tooth surfaces that contain plaque/ The maximum plaque index would be 100%, which represents all surfaces of the patient's teeth containing plaque.
O'Leary Index of Plaque Control | At hygiene appointment (present day) and retrospectively from the clinical record from first hygiene appointment at clinic, up to 17 years previously
  The patient's plaque index= the number of plaque-containing surfaces divided by the total number of available surfaces. The minimum plaque index would be 0% which represents no tooth surfaces that contain plaque/ The maximum plaque index would be 100%, which represents all surfaces of the patient's teeth containing plaque.
Tooth loss | Pre-sanative therapy
  Will be measured as the number of teeth lost due to periodontal disease
Tooth loss | 8-12 weeks post-sanative therapy
  Will be measured as the number of teeth lost due to periodontal disease
Tooth loss | At maintenance appointment (present day) and retrospectively from the clinical record from first maintenance appointment after the 8-12 weeks post-sanative therapy
  Will be measured as the number of teeth lost due to periodontal disease
Tooth loss | At hygiene appointment (present day) and retrospectively from the clinical record from first hygiene appointment at clinic, up to 17 years previously
  Will be measured as the number of teeth lost due to periodontal disease

CONTACTS AND LOCATIONS:
Overall Officials: Wendy E Ward, PhD, Principal Investigator — Brock University
Locations (1):
- Dr. Peter C. Fritz, Periodontal Wellness & Implant Surgery, Fonthill, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Undecided